CLINICAL TRIAL: NCT05861401
Title: Polymorphism of Janus Kinase 1 and 2 (JAK 1&2) in Patients With Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Susanna Fayez Fanos, Resident of dermatology and venerology and Andrology Department-El baliana Genral Hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-23-04-08MS
Record Dates: First submitted 2023-05-03; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Janus Kinase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Under complete sterile precautions, 3mL of blood will be withdrawn by venipuncture and put in EDTA tube; DNA extraction will be done after centrifugation and used for genotyping assay of (JAK 1 and JAK2) gene with the polymerase chain reaction(PCR).
  Interventions: Genetic: Janus Kinase 1 and 2
- cases (Active Comparator): Under complete sterile precautions, 3mL of blood will be withdrawn by venipuncture and put in EDTA tube; DNA extraction will be done after centrifugation and used for genotyping assay of (JAK 1 and JAK2) gene with the polymerase chain reaction(PCR).
  Interventions: Genetic: Janus Kinase 1 and 2

INTERVENTIONS:
Genetic: Janus Kinase 1 and 2 — Under complete sterile precautions, 3mL of blood will be withdrawn by venipuncture and put in EDTA tube; DNA extraction will be done after centrifugation and used for genotyping assay of (JAK 1 and JAK2) gene with the polymerase chain reaction(PCR).

SUMMARY:
Introduction Alopecia areata (AA) is a complex inflammatory disease characterized by cellular infiltration of T- lymphocytes targeting hair follicles, disrupting the anagen phase, with spontaneous remission, recurrence, and exacerbation, making it very unpredictable and emotionally disturbing . It affects nearly 1-2% of the general population with a lifetime risk of 2%, The onset of AA might be at any age; however, most patients develop the disease before 40 years of age . Early-onset AA (a mean age of onset at 5-10 years) predominantly presents as a more severe subtype, such as alopecia universalis . Alopecia areata presents clinically as a non-scarring patchy hair loss primarily on the scalp, and/or other hairy areas and may progress to total scalp hair loss (alopecia totalis, AT ) or complete body hair loss (alopecia universalis, AU ) . Approximately 5- 10% of AA patients will progress into AT/AU . The course of AA varies greatly, the strongest predictors of a poor prognosis include AT, AU, or ophiasis pattern hair loss, as well as earlier age of onset . Severe and recurrent AA disturbs quality of life of patients and may also lead to depression, changed self-image,and interferes with social activities . Currently, the hypotheses for AA development mostly focus on the collapse of immune privilege properties of the hair follicles(HFs) and the nature of self-antigen presentation (follicular antigens) that result in the induction and subsequent attack of activated lymphocytes . Activation of the lymphocytes mainly CD8+NKG2D+induces release of severalTh1 cytokines; interleukin (IL)-1α , IL-1β , and tumor necrosis factor (TNF) alpha, capable of inhibiting (HF) growth with early termination of anagen . AA is a polygenic disorder in which several major genes dictate susceptibility to disease, up to 28% of patients report at least one affected family member, monozygotic twins have exhibited similar times of onset and patterns of hair loss.

Genes loci for Human leucocyte antigens (HLA)DRB1* 1104 and DQB1* 03 are detected in patients with AA. The Janus kinases (JAKs) and signal transducer and activator of transcription (STAT); (JAK/STAT) pathway play an important role in inflammatory processes as they are involved in signaling for over 50 cytokines and growth factors. The JAK/STAT pathway transduces multiple extracellular signals involved in cell proliferation, differentiation, migration, and apoptosis .

The JAK family is constituted by four types of cytoplasmic tyrosine kinases:

JAK1, JAK2, JAK3, and TYK2 . STAT, of which there are seven different subtypes (STAT1, STAT2, STAT3, STAT4, STAT5a, STAT5b, and STAT6) (17), is the other fundamental component of the cascade . After being phosphorylated by JAK, STAT translocates to the nucleus to induce the transcription of specific genes. Alterations in the JAK/STAT pathway have been related to the pathophysiology of atopic dermatitis (AD), vitiligo, and AA.

ELIGIBILITY:
Inclusion Criteria:

* All types of AA.

Exclusion Criteria:

* 1. Pregnancy . 2. Lactation . 3. Systemic diseases . 4. Dermatological disease as vitiligo , psoriasis , atopy . 5. Patient on skin medication affect hair growth as chemotherapy , antithyroid drugs .

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
janus kinase 1 and 2 (JAK 1&2) polymorphism is a risk factor for development of alopecia areata . | 12 months
  different janus kinase 1 and 2 (JAK 1&2) genotypes in alopecia areata in comparison to healthy control.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirzoyev SA, Schrum AG, Davis MDP, Torgerson RR. Lifetime incidence risk of alopecia areata estimated at 2.1% by Rochester Epidemiology Project, 1990-2009. J Invest Dermatol. 2014 Apr;134(4):1141-1142. doi: 10.1038/jid.2013.464. Epub 2013 Nov 11. No abstract available. PMID 24202232
- [Background] Alkhalifah A, Alsantali A, Wang E, McElwee KJ, Shapiro J. Alopecia areata update: part I. Clinical picture, histopathology, and pathogenesis. J Am Acad Dermatol. 2010 Feb;62(2):177-88, quiz 189-90. doi: 10.1016/j.jaad.2009.10.032. PMID 20115945
- [Background] Gilhar A, Kalish RS. Alopecia areata: a tissue specific autoimmune disease of the hair follicle. Autoimmun Rev. 2006 Jan;5(1):64-9. doi: 10.1016/j.autrev.2005.07.001. Epub 2005 Aug 8. PMID 16338213
- [Background] Shapiro J. Clinical practice. Hair loss in women. N Engl J Med. 2007 Oct 18;357(16):1620-30. doi: 10.1056/NEJMcp072110. No abstract available. PMID 17942874